CLINICAL TRIAL: NCT04330027
Title: Effectiveness of Lyophilized Growth Factors for Subacromial Impingement: Randomized Double Blind Placebo Controlled Study
Brief Title: Effectiveness of Lyophilized Growth Factors for Subacromial Impingement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0106178
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-03

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Intercellular Signaling Peptides and Proteins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth factors (Experimental): Patients in this group will receive one lyophilized Growth Factors injection supplied as a powder in a tightly sealed container.
  Interventions: Biological: Growth factors
- Saline (Placebo Comparator): Patients in this group will receive an injection with equal volume of saline; i.e 2ml of 0.9% sodium chloride.
  Interventions: Other: Saline

INTERVENTIONS:
Biological: Growth factors — A new patented product named lyophilized Growth Factors that is an advanced and refined form of conventional platelet-rich plasma
  Arms: Growth factors
Other: Saline — 0.9% Sodium Chloride
  Arms: Saline

SUMMARY:
The aim of this study is to evaluate the efficacy of ultrasound-guided injection of platelet-derived lyophilized growth factors in treatment of subacromial impingement.

DETAILED DESCRIPTION:
A new patented product named lyophilized Growth Factors has been developed. It is a novel advanced and refined form of conventional platelet-rich plasma. Effectiveness of intra-articular lyophilized Growth Factors injection has been studied in thirty patients with symptomatic primary knee osteoarthritis and has shown encouraging results regarding improvement of pain, stiffness and function in addition to decreasing knee effusion.

The lack of good quality evidence to support the efficacy of injecting platelet-derived lyophilized growth factors in treatment of subacromial impingement highlights the need for thorough evaluation of the outcome of this novel therapeutic option in patients with subacromial impingement.

ELIGIBILITY:
Inclusion Criteria:

* Clinically:

  1. Anterolateral shoulder and/or lateral upper arm pain.
  2. Painful arc of motion between 70° and 120°.
  3. Positive impingement sign (Neer's test or Hawkins-Kennedy test).
* Ultrasonographically:

The elicitation of a transient arc of pain during shoulder abduction which coincides with passage of the supraspinatus insertion beneath the coraco-acromial arch.

Exclusion Criteria:

* History of shoulder surgery, fracture, dislocation or subluxation.
* Patients with full-thickness rotator cuff tear, weakness on arm elevation, or positive "drop arm sign".
* Patients who have been diagnosed with a frozen shoulder or degenerative arthropathy of the glenohumeral joint.
* Patients with disorders of the cervical spine or upper extremity that have a significant impact on the shoulder
* Patients with diabetes mellitus, rheumatoid arthritis, hypothyroidism or other painful or function limiting disorders of the shoulder.
* Significant cardiovascular, renal or hepatic disease.
* Active infection in the area to be treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
VAS (Visual Analogue Scale) | 8 weeks
  Pain assessment scale. The minimum value is zero and the maximum value is 10. A higher score indicates a worse outcome.
SPADI (Shoulder Pain and Disability Index) | 8 weeks
  An index measuring the impact of shoulder pathology in terms of pain and disability.
  Total pain score: / 50 x 100 = % Total disability score: / 80 x 100 = % Total Spadi score: / 130 x 100 = % (Note: If a person does not answer all questions divide by the total possible score, eg. if 1 question missed divide by 120) The means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst).
  A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jailan Noureldin, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University Hospitals, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Sherif SM, Abdel-Hamid MM, Noureldin JMAM, Fahmy HM, Abdel-Naby HMA. Effectiveness of lyophilized growth factors injection for subacromial impingement syndrome: a prospective randomized double-blind placebo-controlled study. J Orthop Surg Res. 2023 Jan 31;18(1):78. doi: 10.1186/s13018-023-03548-4. PMID 36721157